CLINICAL TRIAL: NCT04707274
Title: Reliability, Validity, and Cross-cultural Adaptation of the Turkish Version of the Victorian Institute of Sports Assessment for Gluteal Tendinopathy (VISA-G) Questionnaire
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Other Study IDs: E.137836
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2022-01

CONDITIONS: Greater Trochanteric Pain Syndrome of Both Lower Limbs; Gluteal Tendinitis
Keywords: Validity; Reliability; Greater Trochanteric Pain Syndrome; Gluteal tendinopathy
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients group: Individuals with greater trochanteric pain syndrome and gluteal tendinopathy
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Victorian Institute of Sports Assessment for Gluteal Tendinopathy (VISA-G) Questionnaire will be applied.

SUMMARY:
The purpose of this study was to investigate adaptation, validity, and reliability of the Turkish version of the Victorian Institute of Sports Assessment for Gluteal Tendinopathy (VISA-G) Questionnaire.

DETAILED DESCRIPTION:
Gluteal tendinopathy, also known as greater trochanteric pain syndrome, interferes with physical function and sleep, and is characterized by pain and tenderness over the greater trochanter.Clinical risk factors for the development of this condition include advanced age, female gender, back pain, overweight / obesity, poor abductor hip function, altered gait parameters, and psychological distress. The Victorian Institute of Sports Assessment for Gluteal tendinopathy (VISA-G) Questionnaire has recently designed as a patient-reported condition-specific outcome measurement tool to assess disability due to tendinopathy. VISA-G is scored between 0 and 100 (a higher score is expected) and consists of eight items covering three main areas (pain, function, and current activity level). Visual analog score for pain (0-10), the effect of pain on weight-bearing activities (0-30), and difficulty and / or function-related stairs use, including lying on the symptomatic side (0-10), climbing ramps (0-10), standing up without sitting (0-10), home or garden work (0-10) and regular exercise (0-10), physical activity and sports participation (0-10) are evaluated. The study is planned with 40 individuals with gluteal tendinopathy. After questioning the sociodemographic characteristics of the individuals, the patients will be asked to fill in VISA-G, Short Form-36, International Physical Activity Questionnaire, Numeric Rating Scale, Oswestry Disability Index, Oxford Hip Score and modified Harris Hip Score.Test-retest will be re-applied to those of the same individuals who can be reached after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Trochanteric bursitis and/or gluteal tendinopathy,
* Lateral hip pain,
* Pain on palpation of the greater trochanter,
* History of pain when lying on the ipsilateral side or during weight-bearing activities, aggravated by activity for more than 3 months.

Exclusion Criteria:

* Hip osteoarthritis,
* Systemic inflammatory disease such as rheumatoid arthritis,
* Lumbar spine nerve root findings,
* History of lumbar spine or ipsilateral hip joint surgery,
* Osteogenic disease such as Paget's disease,
* Corticosteroid injection to the ipsilateral hip in the past 3 months,
* Hip surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with diagnosis of greater trochanteric pain syndrome and gluteal tendinopathy.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment for Gluteal Tendinopathy (VISA-G) Questionnaire | 10 minutes
  Victorian Institute of Sports Assessment for Gluteal Tendinopathy Questionnaire is designed to assess disability due to gluteal tendinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Seyit CITAKER, Dr., Principal Investigator — Gazi University, Faculty of Health Sciences; M. Baybars ATAOGLU, Dr., Principal Investigator — Gazi University, Faculty of Medicine; Gokhan MARAS, MSc., Principal Investigator — Gazi University, Faculty of Health Sciences; Halime ARIKAN, MSc., Principal Investigator — Ankara University, Faculty of Health Sciences; I. Hazal AYAS, MSc., Principal Investigator — Gazi University, Faculty of Health Sciences; Beyza YAZGAN DAGLI, MSc., Principal Investigator — Gazi University, Faculty of Health Sciences
Locations (1):
- Halime ARIKAN, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR